CLINICAL TRIAL: NCT03172260
Title: An Observational Clinical Trial to Examine the Improvement of E Balance Pro Therapy on Diabetes and Related Complications
Brief Title: Effect of E Balance Pro Therapy on Diabetes and Related Complications
Status: Completed | Type: Observational
Sponsor: CellMedX Corporation (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Other Study IDs: CELLRPD-160001-RPD00
Record Dates: First submitted 2017-05-05; First posted 2017-06-01 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: E Balance Pro Therapy — Micro-current treatment

SUMMARY:
This is an observational study, to test the hypothesis that E Balance Pro Therapy micro-current treatments, delivered with precision in amplitude, waveform and pulsing pattern, adapted by other aspects of this device's technology could affect ion flow across cells and tissues in a fashion that modifies or transforms a crucial pathophysiologic deficit present in patients with diabetes. E Balance Pro Therapy can supplement standard treatment, as an adjunct, and help patients better manage their diabetes. HbA1C is the primary endpoint of this study. However, we expect to see changes in other symptoms (if present) associated with diabetes such as: blood pressure, insulin sensitivity, neuropathic pain retinopathy and wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults > 18 years of age.
* HbA1c 7.0% to 11.0% (inclusive).
* Body mass index 40.0kg/m2 or less.
* Non-smoker, or ex-smoker ≥3 months.
* Female participants of childbearing potential [i.e. not surgically sterilized or post-menopausal (greater than one year since last menses)] must have negative urine pregnancy test and must be using an effective birth control method, defined as:

  * Continuous use of oral or long acting injected contraceptive for at least 2 months prior to study entry, or
  * Use of an intra-uterine device or implantable contraceptive, or
  * Use of double barrier methods of birth control, or
  * Abstinence from heterosexual intercourse.
* Currently on lifestyle management and/or standard treatment for diabetes.
* Currently under the care of a physician.
* Able and willing to perform self-monitoring of plasma glucose regularly.
* Willing to avoid alcohol consumption for 24 h prior to every clinic visit.
* Willing to maintain a stable body weight, activity level, and dietary pattern, except for use of the study products, as directed.
* Willing and able to provide informed written consent prior to any study procedures.

Exclusion Criteria:

* Pregnancy or lactation, or participant unwilling to take appropriate contraceptives for the duration of the study
* History of significant cardiovascular or coronary heart disease (CVD or CHD) as defined by having had a coronary artery bypass procedure, coronary stent or angioplasty, or myocardial infarction in the past six (6) months.
* Current or recent (within six month of Visit 1) history of significant gastrointestinal, renal, pulmonary, hepatic or biliary disease, other endocrine diseases or invasive weight loss treatment.
* Subjects currently using pacemakers.
* History of epilepsy.
* Uncontrolled hypertension (blood pressure SBP > 180 and/or DBP ≥ 105 mm Hg) and unstable use (i.e. initiation or change in dose) of antihypertensive medications or thyroid hormone replacement medications within 3 months prior to Visit 1.
* Plasma creatinine above 130µmol/L or ALT more than twice (2x) upper limit of normal.
* Use of anticoagulants such as (not exhaustive):warfarin (Coumadin), dabigatran (Pradaxa), apixaban (Eliquis) or rivaroxaban (Xarelto). NOTE: Anti-platelet agents such as Plavix are allowed.
* Use of prescription non-steroidal anti-inflammatory drugs (or daily use of over the counter non-steroidal anti-inflammatory drugs >1month), steroids, corticosteroids, or any other prescription anti-inflammatory drugs within three (3) months prior to Visit 1.
* Use of any weight-loss programs or weight-loss medications (prescription or over- the counter) including, but not limited to, lipase inhibitors, within three (3) months prior to Visit 1.
* History of cancer (excluding non-melanoma skin cancer and basal cell carcinoma) in the past five (5) years.
* Presence or history (past 6 months) of alcohol or drug abuse; alcohol use of >2 standard alcoholic drinks per day (one drink= 12oz. beer, 4 oz. wine, 1.5 oz. hard liquor).
* Subject planning to undergo surgery during the study period or up to one (1) month after the study.
* Participant has a known allergy or intolerance to the test products or placebo.
* Participant is unwilling or unable to abide by the requirements of the protocol.
* Any condition that would interfere with the participant's ability to comply with study instructions, might confound the interpretation of the study, or put the participant at risk
* Participant has taken an investigational health product or has participated in a research study within 30 days prior to first study visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a diagnosis of Type 1 or Type 2 Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
HbA1c | 3 months
  change from baseline

SECONDARY OUTCOMES:
Kidney function | 3 months
  Change in serum creatinine from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Hamilton Medical Research Group, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No